CLINICAL TRIAL: NCT04578912
Title: Transcranial Magnetic Stimulation to Augment Behavior Therapy for Tics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSYCH-2020-29064
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Tic Disorders; Tics; Tic, Motor; Tic Disorder, Childhood; Tourette Syndrome; Tourette Syndrome in Children; Tourette Syndrome in Adolescence
MeSH Terms: conditions — Tic Disorders; Tics; Tourette Syndrome | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- CBIT + rTMS (Active Comparator): Participants in this arm will receive Comprehensive Behavioral Intervention for Tics (CBIT) with 1 Hz repetitive Transcranial Magnetic Stimulation (rTMS).
  Interventions: Behavioral: Comprehensive Behavioral Intervention for Tics (CBIT); Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- CBIT + cTBS (Active Comparator): Participants in this arm will receive Comprehensive Behavioral Intervention for Tics (CBIT) with continuous Theta Burst Stimulation (cTBS).
  Interventions: Behavioral: Comprehensive Behavioral Intervention for Tics (CBIT); Device: Continuous Theta Burst Stimulation (cTBS)
- CBIT + Sham (Sham Comparator): Participants in this arm will receive Comprehensive Behavioral Intervention for Tics (CBIT) with either a cTBS or rTMS sham treatment.
  Interventions: Behavioral: Comprehensive Behavioral Intervention for Tics (CBIT)

INTERVENTIONS:
Behavioral: Comprehensive Behavioral Intervention for Tics (CBIT) — CBIT is a manualized treatment program focused on tic management skills
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — During repetitive transcranial magnetic stimulation (rTMS), a electromagnetic coil is placed against the scalp while an electromagnet painlessly delivers a magnetic pulse that stimulates nerve cells in the target brain region
  Arms: CBIT + rTMS
Device: Continuous Theta Burst Stimulation (cTBS) — During continuous theta burst stimulation (cTBS), a electromagnetic coil is placed against the while an electromagnet painlessly delivers magnetic bursts that stimulate nerve cells in the target brain region
  Arms: CBIT + cTBS

SUMMARY:
The study will examine whether combining Comprehensive Behavioral Intervention for Tics (CBIT) with inhibition of the supplementary motor area (SMA) using transcranial magnetic stimulation (TMS) normalizes activity in the SMA-connected circuits, improves tic suppression ability, and enhances CBIT outcomes in young people with tic disorder. The study will also examine different TMS dosing strategies.

DETAILED DESCRIPTION:
All participants will receive 10 daily sessions of CBIT, a well-established behavioral treatment that is considered by the American Academy of Neurology to be the first-line intervention for tics. Immediately prior to each CBIT session, participants will undergo TMS targeting the SMA. The specific type of TMS procedure will be randomly assigned between subjects and be either: 1 Hz repetitive TMS (rTMS), continuous theta burst stimulation (cTBS), or sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Current chronic motor and/or vocal tics, defined as tics for at least 1 year without a tic-free period of more than 3 consecutive months. Tics must not be due to a medical condition or the direct physiological effects of a substance.
* At least moderate tic severity, defined as a Yale Global Tic Severity Scale total score ≥14 (≥9 for those with motor or vocal tics only).
* Full scale IQ greater than or equal to 70
* English fluency to ensure comprehension of study measures and instructions.
* Right-handed

Exclusion Criteria:

* Medical conditions contraindicated or associated with altered TMS risk profile, including history of intracranial pathology, epilepsy or seizure disorders, traumatic brain injury, brain tumor, stroke, implanted medical devices or metallic objects in the head, current pregnancy or participants of childbearing age not using effective contraception, or any other medical condition deemed serious or contraindicated by a study physician
* Inability to undergo MRI.
* Left handedness.
* Active suicidality.
* Previous diagnosis of psychosis or cognitive disability.
* Substance abuse or dependence within the past year.
* Concurrent psychotherapy focused on tics.
* Neuroleptic/antipsychotic medications.
* Taking a medication that has not reached stability criterion (same medication and dose for 6 weeks with no planned changes over the intervention period)

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Conelea, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Some datasets (to be determined) will be made available via NIH National Database Archive.

REFERENCES:
- [Derived] Conelea C, Greene DJ, Alexander J, Houlihan K, Hodapp S, Wellen B, Francis S, Mueller B, Hendrickson T, Tseng A, Chen M, Fiecas M, Lim K, Opitz A, Jacob S. The CBIT + TMS trial: study protocol for a two-phase randomized controlled trial testing neuromodulation to augment behavior therapy for youth with chronic tics. Trials. 2023 Jul 3;24(1):439. doi: 10.1186/s13063-023-07455-1. PMID 37400828
- [Derived] Conelea C, Greene D, Alexander J, Houlihan K, Hodapp S, Wellen B, Francis S, Mueller B, Hendrickson T, Tseng A, Chen M, Fiecas M, Lim K, Opitz A, Jacob S. The CBIT+TMS Trial: study protocol for a two-phase randomized controlled trial testing neuromodulation to augment behavior therapy for youth with chronic tics. Res Sq [Preprint]. 2023 Jun 13:rs.3.rs-2949388. doi: 10.21203/rs.3.rs-2949388/v1. PMID 37398344

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator: 1 Hz rTMS: Participants in this arm will receive Comprehensive Behavioral Intervention for Tics (CBIT) with 1 Hz repetitive Transcranial Magnetic Stimulation (rTMS).
- Active Comparator: cTBS: Participants in this arm will receive Comprehensive Behavioral Intervention for Tics (CBIT) with continuous Theta Burst Stimulation (cTBS).
- Sham Comparator: Sham: Participants in this arm will receive Comprehensive Behavioral Intervention for Tics (CBIT) with sham stimulation.
Period: Overall Study
Arm/Group | Active Comparator: 1 Hz rTMS | Active Comparator: cTBS | Sham Comparator: Sham
Started | 17 | 16 | 17
Completed | 17 | 15 | 16
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator: 1 Hz rTMS | Active Comparator: cTBS | Sham Comparator: Sham | Total
Number analyzed (Participants) | 17 | 16 | 17 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 12 | 12 | 37
  Between 18 and 65 years | 4 | 4 | 5 | 13
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 7 | 23
  Male | 9 | 8 | 10 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 13 | 14 | 15 | 42
  More than one race | 2 | 2 | 2 | 6
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Resting State fMRI Connectivity of SMA-mediated Brain Circuits
Description: For each participant, signal intensity (unitless measure) will be measured using fMRI in the supplementary motor area (SMA) during a finger tapping task. An ANOVA will be conducted to compare change in signal intensity within SMA from pre- to post-treatment across the groups. The outcome will be reported as an effect size value (Cohen's d).
Time Frame: baseline to post-treatment; approximately 10 days
Measure: Mean (Standard Deviation); unit: eta squared
Arm/Group | CBIT + rTMS | CBIT + cTBS | CBIT + Sham
Number analyzed (Participants) | 15 | 13 | 17
eta squared | 0.0312 (0.05) | 0.261 (0.05) | 0.158 (0.03)

2. Primary Outcome: Change in SMA Activation
Description: as for outcome 1
Time Frame: baseline to post-treatment; approximately 10 days
Measure: Mean (Standard Deviation); unit: eta squared
Arm/Group | CBIT + rTMS | CBIT + cTBS | CBIT + Sham
Number analyzed (Participants) | 15 | 13 | 17
eta squared | 0.45 (1.25) | 0.01 (1.25) | 0.27 (1.3)

3. Secondary Outcome: Safety: Measured as Rate of Adverse Events Related to Study Treatment
Description: The number of adverse events judged to be treatment related will be totaled and reported for each group.
Time Frame: approximately 3-4 months
Measure: Number; unit: events
Arm/Group | CBIT + rTMS | CBIT + cTBS | CBIT + Sham
Number analyzed (Participants) | 17 | 16 | 17
events | 46 | 22 | 18

4. Secondary Outcome: Change in Tic Suppression Task
Description: The Tic Suppression Task is a clinician-rated tool for assessing tic frequency. A video recording of participant is rated and yields a score in units of tics per minute. Outcome reported as change from baseline to post treatment; change from baseline to 1 month post treatment; change from baseline to 3 months post treatment; change from post treatment to 1 month post treatment; and change from post treatment to 3 months post treatment.
Time Frame: baseline to 3 months post-treatment
Measure: Mean (Standard Deviation); unit: tics per minute
Arm/Group | CBIT + rTMS | CBIT + cTBS | CBIT + Sham
Number analyzed (Participants) | 17 | 16 | 17
tics per minute | 0.58 (9.47) | -3.83 (23.92) | -8.24 (15.71)

5. Secondary Outcome: Feasibility: Measured as Participant Treatment Completion
Description: For each group, the number of participants who completed at least 80% of treatment sessions will be totaled and reported for each group.
Time Frame: approximately 3-4 months
Measure: Number; unit: participants
Arm/Group | CBIT + rTMS | CBIT + cTBS | CBIT + Sham
Number analyzed (Participants) | 17 | 16 | 17
participants | 17 | 15 | 16

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Active Comparator: 1 Hz rTMS | Active Comparator: cTBS | Sham Comparator: Sham
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 17/17 | 15/15 | 14/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: 1 Hz rTMS (N=17) | Active Comparator: cTBS (N=15) | Sham Comparator: Sham (N=16)
Headache (General disorders) | 7 (21) | 6 (10) | 7 (9)
Muscle Twitch (Musculoskeletal and connective tissue disorders) | 7 (8) | 0 (0) | 2 (2)
sleep disturbance (General disorders) | 4 (5) | 3 (3) | 1 (1)
Other (General disorders) | 2 (2) | 1 (1) | 2 (4)
Mood change (General disorders) | 2 (4) | 1 (2) | 0 (0)
Pain (General disorders) | 1 (2) | 1 (2) | 2 (2)
Nausea (General disorders) | 1 (1) | 1 (2) | 0 (0)
Scalp discomfort (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Concentration difficulties (General disorders) | 1 (1) | 1 (1) | 0 (0)
Hearing difficulties (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/12/NCT04578912/Prot_SAP_002.pdf
  • Informed Consent Form (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT04578912/ICF_001.pdf